CLINICAL TRIAL: NCT02709707
Title: A Lay User Study of the iGlucose, a Device for Self-Monitoring of Blood Glucose (SMBG), Marketed by the Smart Meter Corporation
Brief Title: Lay-user Trial of the iGlucose Blood Glucose Monitoring System
Status: Completed | Type: Observational
Sponsor: Nina Peled (Industry)
Responsible Party: Sponsor-Investigator, Nina Peled, Regulatory Consultant, Smart Meter Corporation
Organization: Smart Meter Corporation (Industry)
Other Study IDs: CP00001
Record Dates: First submitted 2016-03-08; First posted 2016-03-16 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-06

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes, Blood Sugar
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with diabetes
  Interventions: Device: Blood glucose monitor

INTERVENTIONS:
Device: Blood glucose monitor

SUMMARY:
Evaluation of the iGlucose Blood Glucose Monitoring System in the hands of lay users

DETAILED DESCRIPTION:
A non-randomized, prospective study of recruited subjects with diabetes. Subjects will include those with type I or type II diabetes of various duration and those who are naive to self-testing of blood glucose. Subjects will use provided instructions-for-use to undergo self-training on the use of the device and will then self-test their blood glucose level. Results will be compared to those obtained by a lab glucose analyzer.

ELIGIBILITY:
Inclusion Criteria:

* Be 12 years of age and older
* Have pre-existing diagnosis of diabetes
* Be able to read and understand English
* Agree to participate in the study
* Be able and willing to provide informed consent

Exclusion Criteria:

* Do not meet Inclusion Criteria
* With Hemophilia or any other bleeding disorder
* With any condition which in the opinion of the Investigator may place the subject or site staff at excessive risk
* With physical condition/limitation preventing the use of SMBG on their own

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with a diagnosis of diabetes, either type 1 or type 2, of various duration with blood glucose levels covering the entire measurement range. .
Sampling Method: Non-Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2016-03; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Accuracy of blood glucose measurements as performed by lay users | 10 minutes to produce self blood result and to perform lab comparative method

SECONDARY OUTCOMES:
Assessment by lay users of the ease of use of the iGlucose Blood Glucose Monitoring System | 2 -3 hours of going through a self-training session and producing an assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Diablo Clinical Research, Walnut Creek, California, United States

IPD SHARING:
Plan to Share IPD: No